CLINICAL TRIAL: NCT01886248
Title: Antithrombin-III for Patients With Hepatic Veno-occlusive Diseases Following Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Antithrombin-III
Record Dates: First submitted 2013-05-30; First posted 2013-06-25 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Hepatic Veno-Occlusive Disease
Keywords: hepatic veno-occlusive disease after hematopoietic stem cell transplantation
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease | interventions — Antithrombin III

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antithrombin-III Human 500IU (Experimental): Freeze-dried Concentrated Human Antithrombin Ⅲ 500 IU
  Units required (IU)/kg = 50 + [(desired-baseline AT-III level) x weight (kg) / 1.4]
  Interventions: Drug: Freeze-dried Concentrated Human Antithrombin Ⅲ 500 IU

INTERVENTIONS:
Drug: Freeze-dried Concentrated Human Antithrombin Ⅲ 500 IU
  Other Names: Antithrombin-III Human 500IU

SUMMARY:
To evaluate efficacy and safety of AT-III treatment in patients with hepatic veno-occlusive diseases following hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hepatic veno-occlusive disease after hematopoietic stem cell transplantation. The following criteria will be used.

   1. Two of the following

      * Serum total bilirubin > 2.0 mg/dL
      * Hepatomegaly or right upper quadrant pain of liver origin
      * Unexplained weight gain of>2% over baseline because of fluid accumulation
   2. Patients with pathologic diagnosis.
2. Patients with informed consent

Exclusion Criteria:

1. Pregnant or nursing women.
2. Malignant or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
3. Psychiatric disorder that would preclude compliance.
4. Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
5. History of anaphylactic reaction to the study drug

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-06; Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
AT-III level before 5th dose of AT-III | up to 14 days

SECONDARY OUTCOMES:
AT-III level before 9th dose | up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, MD, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Chongno-gu, South Korea